CLINICAL TRIAL: NCT04866121
Title: The Comparison of P6+ST36 Combination Acupuncture Therapy With P6 Alone Acupuncture and Standard Treatment in Postoperative Nausea and Vomiting
Brief Title: Acupuncture for Prevention of Postoperative Nausea and Vomiting
Acronym: PONV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Alirıza Erdoğan, Principal Investigator, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14.04.2021/28
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: PONV
Keywords: PONV; P6 Acupuncture; ST36 Acupuncture
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Treatment (No Intervention): Following 8 hours fasting, standard anesthesia protocol, 3 mg kg-1 Propofol, 0.6 mg kg-1 rocuronium and 2 µg kg-1 fentanyl will be administered. Laparoscopic cholecystectomy will be performed. Twenty minutes prior to the completion of the operation tramadol 100mg will be administered for analgesia.
- Single point (P6) Acupuncture (Active Comparator): Prior to the anesthesia induction, the same certified medical doctor will perform a standard acupuncture protocol to the P6 point bilaterally. For P6 acupuncture stimulation 0,25x25mm steel needles will be immersed for 2cm. For stimulation, the needles will be turned clock-wise 3 times. This stimulation will be repeated for 3 times with 10 seconds intervals. The needles will be held in place for 20 minutes and will be removed afterwards.
  Following 8 hours fasting, standard anesthesia protocol, 3 mg kg-1 Propofol, 0.6 mg kg-1 rocuronium and 2 µg kg-1 fentanyl will be administered. Laparoscopic cholecystectomy will be performed. Twenty minutes prior to the completion of the operation tramadol 100mg will be administered for analgesia.
  Interventions: Procedure: Acupuncture
- Double point (P6+ST36) Acupuncture (Experimental): Prior to the anesthesia induction, the same certified medical doctor will perform a standard acupuncture protocol both to the P6 and ST36 points bilaterally. For P6 acupuncture stimulation 0,25x25mm steel needles will be immersed for 2cm. For ST6 acupuncture stimulation 0,25x50mm steel needles will be immersed for 5cm. For stimulation, the needles will be turned clock-wise 3 times. This stimulation will be repeated for 3 times with 10 seconds intervals. The needles will be held in place for 20 minutes and will be removed afterwards. Following 8 hours fasting, standard anesthesia protocol, 3 mg kg-1 Propofol, 0.6 mg kg-1 rocuronium and 2 µg kg-1 fentanyl will be administered. Laparoscopic cholecystectomy will be performed. Twenty minutes prior to the completion of the operation tramadol 100mg will be administered for analgesia.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — A standardized acupuncture protocol will be administered
  Arms: Double point (P6+ST36) Acupuncture; Single point (P6) Acupuncture

SUMMARY:
The aim of this study is to compare the single point stimulation (P6) and double point stimulation (P6+ST36) performed before anesthesia induction with standard treatment in terms of PONV development and postoperative anti-emetic requirement in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is encountered in 20-30% of patients undergoing surgery. PONV is a costly medical condition in financial and emotional aspects by causing serious complications like elongation of hospital stay, postoperative bleeding, aspiration pneumonia and electrolyte imbalances. In high risk individuals and operations, it can be encountered in up to 80% of patients. The risk factors for PONV development in adults are female gender, previous PONV and/or motion sickness, non-smoking and younger age. Additionally, it has been reported that some surgery types, especially, laparoscopic cholecystectomy and gynecologic surgeries along with the anesthetic agent, the duration of anesthesia and postoperative opioid use also have direct effects on PONV development.

According to the 4th consensus guidelines for the management of PONV updated in 2020, in patients with one or more risk factors, a multimodal prophylaxis using a combination of at least 2 of the following methods; 5-HT3 receptor antagonists, corticosteroids, anti-histaminics, dopamine antagonists, propofol anesthesia, NK-1 receptor antagonists, anti-cholinergics and acupuncture.

Following the declaration of acupuncture as an effective treatment option for PONV in 1999 NIH Consensus Conference, studies about this topic gained speed and many high quality randomized controlled clinic studies were performed. In one of the most comprehensive reviews published in 2015, it is stated that stimulation of P6 acupuncture point remarkably reduce the risk of PONV development, significantly decrease the amount of postoperative anti-emetic requirement, provide similar PONV prophylaxis with different pharmacoprophylactic agents (metoclopramide, cyclizine, prochlorperazine, droperidol, ondansetron and dexamethasone) and have similar post-operative anti-emetic requirement with pharmacologic agents. In the same Cochrane analysis, it is clearly stated that studies enrolling groups of sham acupuncture for P6 are redundant and would not go any further than duplicating the available well-established information. In this aspect, the proposed study design is comparison between treatment groups.

PONV has a multifactorial ethology. It has been postulated that it occurs as a result of activation of emetic center in the brain stem by stimulation of various peripheral receptors as well as central receptors including the chemoreceptor trigger zone in the postrema region. Following activation, the response of emetic center for anti-emetic agents is rather weak and consequently this complicates PONV treatment. Acupuncture is a kind of periphery sensory stimulus and has modulatory effects on the emetic center in the brain stem via neuronal pathways. This neural modulation is thought to be the result of communication between cerebellum and insula. As a result of these mechanisms of action, performing acupuncture before the induction of anesthesia provides more effective PONV prophylaxis.

Pharmacologic anti-emetic agents increase treatment costs as well as bear some adverse effects. The clinical condition created by PONV and increasing dissatisfaction due to the adverse effects of the pharmacologic agents urge both patients and clinicians pursuing non-pharmacologic modalities with proven efficiency, like acupuncture.

Therefore, it is essential to develop a standard, simple, effective prophylaxis protocol with high patient compliance and without ad verse effects, especially in patients with high risk for PONV. In the literature various different technique and materials were used for acupuncture stimulation. Unfortunately, a standard is not present for the metal of the needle, the length of the needle, the depth of immersion, the technique of stimulation and in most of the studies these features are not specified at all. Meanwhile, although P6 is the most studied point for PONV, there are encouraging evidence that some other points, like ST36 or LI4, might be incorporated into the PONV protocol. ST36 have potential effects in balancing gastrointestinal motility by modulating gastric motility via vagovagal and sympathetic reflex arches. Moreover, P6 in combination with ST36 has been successful in treatment of hiccups, recently.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18-65 years old, who have ASA scores of I-II-III and who are planned to undergo elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Pregnant women
* Lactating women
* Women with steel hypersensitivity
* Mental retarded patients
* Patients with psychological disorders and neurologic sequel
* Additionally, patients who;
* have nausea/vomiting, consume anti-emetic or emetogenic drugs, alcohol, opioid drugs, glucocorticoid drug and have acupuncture treatment for any reason 72 hours prior to surgery
* have skin reactions at the site of acupuncture application
* had intraoperative gangrenous cholecystitis, gall bladder perforation, malignant pathological outcome
* were admitted to intensive care unite
* had to convert to open surgery will be excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Laparoscopic cholecystectomy is performed far more in women than in men with a ratio of 5:1. Additionally, being women is one of the major risk factors for PONV development.
Enrollment: 105 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
PONV prophylaxis | 12 months
  The frequency of PONV development
Postoperative anti-emetic requirement | 12 months
  The amount of anti-emetic agent administered postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Niğde Ömer Halisdemir University Training and Research Hospital, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Unsal N, Akcaboy ZN, Soyal OB, Akcaboy EY, Mutlu NM, Gogus N. Effectiveness of Intraoperative Laser Acupuncture Combined with Antiemetic Drugs for Prevention of Postoperative Nausea and Vomiting. J Altern Complement Med. 2020 Jan;26(1):67-71. doi: 10.1089/acm.2019.0181. Epub 2019 Oct 3. PMID 31580707
- [Background] Apfel CC, Heidrich FM, Jukar-Rao S, Jalota L, Hornuss C, Whelan RP, Zhang K, Cakmakkaya OS. Evidence-based analysis of risk factors for postoperative nausea and vomiting. Br J Anaesth. 2012 Nov;109(5):742-53. doi: 10.1093/bja/aes276. Epub 2012 Oct 3. PMID 23035051
- [Background] Lee A, Chan SK, Fan LT. Stimulation of the wrist acupuncture point PC6 for preventing postoperative nausea and vomiting. Cochrane Database Syst Rev. 2015 Nov 2;2015(11):CD003281. doi: 10.1002/14651858.CD003281.pub4. PMID 26522652
- [Background] Usichenko TI, Hesse T. Appropriate timing and intensity of PC6 stimulation for the prevention of postoperative nausea and vomiting. Acupunct Med. 2016 Feb;34(1):70-1. doi: 10.1136/acupmed-2015-010926. Epub 2015 Aug 18. No abstract available. PMID 26286527
- [Background] Bai L, Niu X, Liu Z, Chen Z, Wang X, Sun C, Wang Z, Wang S, Cao J, Gan S, Fan G, Huang W, Xu H, Chen S, Tian J, Lao L, Zhang M. The role of insula-cerebellum connection underlying aversive regulation with acupuncture. Mol Pain. 2018 Jan-Dec;14:1744806918783457. doi: 10.1177/1744806918783457. Epub 2018 Jun 19. PMID 29921161
- [Background] Lu MJ, Yu Z, He Y, Yin Y, Xu B. Electroacupuncture at ST36 modulates gastric motility via vagovagal and sympathetic reflexes in rats. World J Gastroenterol. 2019 May 21;25(19):2315-2326. doi: 10.3748/wjg.v25.i19.2315. PMID 31148903
- [Background] Sun ZG, Pi YL, Zhang J, Wang M, Zou J, Wu W. Effect of acupuncture at ST36 on motor cortical excitation and inhibition. Brain Behav. 2019 Sep;9(9):e01370. doi: 10.1002/brb3.1370. Epub 2019 Jul 30. PMID 31359627
- [Background] Xu J, Qu Y, Yue Y, Zhao H, Gao Y, Peng L, Zhang Q. Treatment of persistent hiccups after arthroplasty: effects of acupuncture at PC6, CV12 and ST36. Acupunct Med. 2019 Feb;37(1):72-76. doi: 10.1136/acupmed-2016-011304. Epub 2019 Mar 7. PMID 30843420